CLINICAL TRIAL: NCT01549964
Title: A Multicenter, Randomized, Double-Blind, Placebo- and Active-Controlled, Phase 3 Study to Evaluate the Efficacy and Safety of TAK-875 25 mg and 50 mg Compared to Placebo and Sitagliptin 100 mg When Used in Combination With Metformin in Subjects With Type 2 Diabetes
Brief Title: Comparison of Fasiglifam (TAK-875) to Placebo and Sitagliptin in Combination With Metformin in Participants With Type 2 Diabetes
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to concerns about potential liver safety (See Detailed Description)
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-875_302; 2011-001752-10 (EudraCT Number); U1111-1124-2225 (Registry Identifier: WHO); NMRR-12-446-11314 (Registry Identifier: NMRR (Malaysia))
Record Dates: First submitted 2012-03-06; First posted 2012-03-09 (Estimated); Results first posted 2016-06-02 (Estimated); Last update posted 2016-06-02 (Estimated); Status verified 2016-04

CONDITIONS: Glycemic Control
Keywords: Drug Therapy
MeSH Terms: interventions — TAK-875; Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Fasiglifam (TAK-875) 25 mg (Experimental): Fasiglifam 25 mg, tablets, orally, once daily for a 24-week Treatment Period followed by an optional 80-week extension period for up to 104 weeks of treatment. Sitagliptin placebo-matching tablets, orally, once daily for a 24-week Treatment Period followed by an optional 80-week extension period for up to 104 weeks of treatment. Metformin ≥1500 mg or Maximum Tolerated Dose (MTD) needs to continue at a stable dose.
  Interventions: Drug: Fasiglifam (TAK-875)
- Fasiglifam (TAK-875) 50 mg (Experimental): Fasiglifam 50 mg, tablets, orally, once daily for a 24-week Treatment Period followed by an optional 80-week extension period for up to 104 weeks of treatment. Sitagliptin placebo-matching tablets, orally, once daily for a 24-week Treatment Period followed by an optional 80-week extension period for up to 104 weeks of treatment. Metformin ≥1500 mg or Maximum Tolerated Dose (MTD) needs to continue at a stable dose.
  Interventions: Drug: Fasiglifam (TAK-875)
- Sitagliptin 100 mg (Active Comparator): Sitagliptin 100 mg, tablets, orally, once daily for a 24-week Treatment Period followed by an optional 80-week extension period for up to 104 weeks of treatment. TAK-875 placebo-matching tablets, orally, once daily for a 24-week Treatment Period followed by an optional 80-week extension period for up to 104 weeks of treatment. Metformin ≥1500 mg or Maximum Tolerated Dose (MTD) needs to continue at a stable dose.
  Interventions: Drug: Sitagliptin
- Placebo (Placebo Comparator): Fasiglifam (TAK-875) placebo-matching tablets, orally, once daily for a 24-week Treatment Period followed by an optional 80-week extension period for up to 104 weeks of treatment. Sitagliptin placebo-matching tablets, orally, once daily for a 24-week Treatment Period followed by an optional 80-week extension period for up to 104 weeks of treatment. Metformin ≥1500 mg or Maximum Tolerated Dose (MTD) needs to continue at a stable dose.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fasiglifam (TAK-875) — Fasiglifam (TAK-875) tablets
  Arms: Fasiglifam (TAK-875) 25 mg; Fasiglifam (TAK-875) 50 mg
Drug: Sitagliptin — Sitagliptin tablets
  Other Names: Januvia
  Arms: Sitagliptin 100 mg
Drug: Placebo — Placebo-matching tablets
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of 2 doses of TAK-875 (25 mg and 50 mg), once daily (QD), plus metformin compared to placebo plus metformin and sitagliptin plus metformin on lowering blood sugar.

DETAILED DESCRIPTION:
TAK-875 is being developed at Takeda Development Center, Inc. as an adjunct to diet and exercise to improve glycemic control in participants with Type 2 Diabetes Mellitus (T2DM) whose blood glucose level is inadequately controlled with metformin.

This study will evaluate the efficacy of TAK-875 (25 mg and 50 mg) plus metformin compared to placebo plus metformin and sitagliptin plus metformin on glycemic control as measured by change from baseline in glycosylated hemoglobin (HbA1c) over a 24-week Treatment Period. Participants completing the 24-week Treatment Period may enter an optional 80-week extension period for a total of 104 weeks of treatment.

Due to concerns about potential liver safety, on balance, the benefits of treating patients with fasiglifam (TAK-875) do not outweigh the potential risks.

For this reason, Takeda has decided voluntarily to terminate the development activities for fasiglifam.

ELIGIBILITY:
Inclusion Criteria:

1. The participant is male or female and 18 years of age or older with a historical diagnosis of type II diabetes mellitus.
2. The participant meets one of the following criteria:

   1. The participant has an HbA1c level ≥7.5 and <10.5%, and has been on a stable daily dose of ≥1500 mg (or documented maximum tolerated dose [MTD]) of metformin for at least 2 months prior to Screening. This participant will immediately enter the Placebo Run-in Period according to Study Schedule A, or;
   2. The participant has an HbA1c level ≥7.5 and <10.5%, and has been on a stable daily dose of <1500 mg of metformin without documented MTD for at least 2 months prior to Screening. After completing the Screening Visit, this participant will have their metformin dose immediately increased to ≥1500 mg (or MTD) for an 8-week Titration Period according to Study Schedule B. Following this 8-week period, the participant must qualify for entry into the Placebo Run-in Period by completing the Week -3 procedures including having an HbA1c level ≥7.5 and <10.5%.
3. The participant has had no treatment with antidiabetic agents other than metformin within 2 months prior to Screening (Exception: if a participant has received other antidiabetic therapy for ≤7 days within the 2 months prior to Screening).
4. The participant has a body mass index (BMI) ≤45 kg/m² at Screening.
5. Participants regularly using other, non-excluded medications, must be on a stable dose for at least 4 weeks prior to Screening. However, PRN (as needed) use of prescription or over-the-counter medications is allowed at the discretion of the investigator.
6. The participant is able and willing to monitor glucose with a home glucose monitor and consistently record his or her own blood glucose concentrations and complete subject diaries.

Exclusion Criteria:

1. The participant donated or received any blood products within 12 weeks prior to Screening or is planning to donate blood during the study.
2. Hemoglobin ≤12 g/dL (≤120 g/L) for males and ≤10 g/dL (≤100 g/L) for females at Screening Visit.
3. The participant has systolic blood pressure ≥160 mm Hg or diastolic pressure ≥95 mm Hg at Screening Visit. (If the participant meets this exclusion criterion, the assessment may be repeated once at least 30 minutes after the initial measurement.)
4. The participant has a history of laser treatment for proliferative diabetic retinopathy within 6 months prior to Screening.
5. The participant has had treatment for gastric banding or gastric bypass surgery within one year prior to Screening.
6. The participant had coronary angioplasty, coronary stent placement, coronary bypass surgery, myocardial infarction, unstable angina pectoris, clinically significant abnormal ECG, cerebrovascular accident or transient ischemic attack within 3 months prior to or at Screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 916 (Actual)
Dates: Start 2012-04; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical Director Clinical Science, Study Director — Takeda
Locations (160):
- United States (58):
  - Muscle Shoals, Alabama
  - Mesa, Arizona
  - Peoria, Arizona
  - Phoenix, Arizona
  - Chula Vista, California
  - El Cajon, California
  - La Mesa, California
  - Laguna Hills, California
  - National City, California
  - Paramount, California
  - San Diego, California
  - Stockton, California
  - Tustin, California
  - West Hills, California
  - Trumbull, Connecticut
  - Coral Gables, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - New Port Richey, Florida
  - Ocala, Florida
  - West Palm Beach, Florida
  - Meridian, Idaho
  - Chicago, Illinois
  - Greenfield, Indiana
  - Muncie, Indiana
  - Lexington, Kentucky
  - Owensboro, Kentucky
  - Hyattsville, Maryland
  - Troy, Michigan
  - Picayune, Mississippi
  - St Louis, Missouri
  - Haddon Heights, New Jersey
  - Rosedale, New York
  - Calabash, North Carolina
  - Charlotte, North Carolina
  - Monroe, North Carolina
  - Morehead City, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Dayton, Ohio
  - Norman, Oklahoma
  - Lancaster, Pennsylvania
  - Levittown, Pennsylvania
  - Spartanburg, South Carolina
  - Crossville, Tennessee
  - Memphis, Tennessee
  - Carrollton, Texas
  - Houston, Texas
  - Irving, Texas
  - Katy, Texas
  - McKinney, Texas
  - Plano, Texas
  - San Antonio, Texas
  - Spring, Texas
  - Salt Lake City, Utah
  - West Jordan, Utah
  - Richmond, Virginia
- Australia (8):
  - Camperdown, New South Wales
  - Maroubra, New South Wales
  - Redcliffe, Queensland
  - Adelaide, South Australia
  - Daw Park, South Australia
  - Box Hill, Victoria
  - Fitzroy, Victoria
  - Melbourne, Victoria
- Bulgaria (4):
  - Byala
  - Kazanlak
  - Plovdiv
  - Sofia
- Croatia (8):
  - Čakovec
  - Karlovac
  - Krapinske Toplice
  - Rijeka
  - Slavonski Brod
  - Split
  - Zadar
  - Zagreb
- Czechia (13):
  - Beroun
  - Brno
  - Havlíčkův Brod
  - Kladno
  - Kroměříž
  - Mladá Boleslav
  - Ostrava
  - Ostrava - Moravska Ostrava
  - Pardubice
  - Pilsen
  - Písek
  - Prague
  - Ústí nad Labem
- Hungary (25):
  - Baja
  - Balatonfüred
  - Budaörs
  - Budapest
  - Debrecen
  - Eger
  - Gödöllő
  - Gyöngyös
  - Gyula
  - Hódmezővásárhely
  - Kecskemét
  - Kistelek
  - Kisvárda
  - Komárom
  - Mohács
  - Nyíregyháza
  - Pécs
  - Szeged
  - Szekszárd
  - Szikszó
  - Szolnok
  - Szombathely
  - Úrhida
  - Veszprém
  - Zalaegerszeg
- Italy (4):
  - Florence, Firenze
  - Milan, Milano
  - Sesto San Giovanni, Milano
  - Pavia, Pavia
- Malaysia (8):
  - Johor Bahru, Johor
  - Alor Star, Kedah
  - Kelantan, Kelantan
  - Kota Bharu, Kelantan
  - Cheras, Kuala Lumpur
  - Kuala Lumpur, Kuala Lumpur
  - Lembah Pantai, Kuala Lumpur
  - Petaling Jaya, Selangor
- Slovakia (19):
  - Banská Bystrica
  - Bardejov
  - Bratislava
  - Kosice - Saca
  - Košice
  - Levice
  - Lučenec
  - Moldava nad Bodvou
  - Nitra
  - Pezinok
  - Prešov
  - Prievidza
  - Stropkov
  - Svidník
  - Šahy
  - Štúrovo
  - Trebišov
  - Trenčín
  - Žilina
- South Korea (4):
  - Goyang-si, Gyeonggi-do
  - Seongnam-si, Gyeonggi-do
  - Incheon
  - Seoul
- Thailand (9):
  - Bangkok, Bangkok
  - Patumwan, Bangkok
  - Rachathevi, Bangkok
  - Rajtevi, Bangkok
  - Ratchathewi, Bangkok
  - Khon Kaen, Changwat Khon Kaen
  - Muang, Changwat Nakhon Ratchasima
  - Hat Yai, Changwat Songkhla
  - Muang, Chiang Mai

REFERENCES:
- [Derived] Shavadia JS, Sharma A, Gu X, Neaton J, DeLeve L, Holmes D, Home P, Eckel RH, Watkins PB, Granger CB. Determination of fasiglifam-induced liver toxicity: Insights from the data monitoring committee of the fasiglifam clinical trials program. Clin Trials. 2019 Jun;16(3):253-262. doi: 10.1177/1740774519836766. Epub 2019 Mar 18. PMID 30880443

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 168 investigative sites in Australia, Bulgaria, Croatia, Czech Republic, Hungary, Italy, Korea, Republic, Malaysia, Slovakia, Thailand and the United States from 05 April 2012 to 27 March 2014.
Pre-assignment Details: Participants with a diagnosis of Type 2 Diabetes Mellitus were randomly enrolled in 1 of 4 treatment groups in a 1:2:2:2 ratio, once a day placebo, 100 mg sitagliptin, 25 mg fasiglifam or 50 mg fasiglifam in combination with metformin.
Groups:
- Placebo: Fasiglifam placebo-matching tablets, orally, once daily for a 24-week Treatment Period followed by an optional 80-week extension period for up to 104 weeks of treatment. Sitagliptin placebo-matching tablets, orally, once daily for a 24-week Treatment Period followed by an optional 80-week extension period for up to 104 weeks of treatment. Metformin ≥1500 mg or Maximum Tolerated Dose (MTD) needs to continue at a stable dose.
- Sitagliptin 100 mg: Sitagliptin 100 mg, tablets, orally, once daily for a 24-week Treatment Period followed by an optional 80-week extension period for up to 104 weeks of treatment. Fasiglifam placebo-matching tablets, orally, once daily for a 24-week Treatment Period followed by an optional 80-week extension period for up to 104 weeks of treatment. Metformin ≥1500 mg or Maximum Tolerated Dose (MTD) needs to continue at a stable dose.
- Fasiglifam 25 mg: Fasiglifam 25 mg, tablets, orally, once daily for a 24-week Treatment Period followed by an optional 80-week extension period for up to 104 weeks of treatment. Sitagliptin placebo-matching tablets, orally, once daily for a 24-week Treatment Period followed by an optional 80-week extension period for up to 104 weeks of treatment. Metformin ≥1500 mg or Maximum Tolerated Dose (MTD) needs to continue at a stable dose.
- Fasiglifam 50 mg: Fasiglifam 50 mg, tablets, orally, once daily for a 24-week Treatment Period followed by an optional 80-week extension period for up to 104 weeks of treatment. Sitagliptin placebo-matching tablets, orally, once daily for a 24-week Treatment Period followed by an optional 80-week extension period for up to 104 weeks of treatment. Metformin ≥1500 mg or Maximum Tolerated Dose (MTD) needs to continue at a stable dose.
Period: 24-Week Treatment Period
Arm/Group | Placebo | Sitagliptin 100 mg | Fasiglifam 25 mg | Fasiglifam 50 mg
Started | 132 | 260 | 263 | 261
Safety Analysis Set=Received Treatment | 132 | 260 | 263 | 260
Completed | 71 | 149 | 147 | 140
Not Completed | 61 | 111 | 116 | 121
Not completed — Study Terminated by Sponsor | 50 | 104 | 104 | 105
Not completed — Voluntary Withdrawal | 6 | 3 | 3 | 8
Not completed — Pretreatment Event/Adverse Event | 1 | 4 | 4 | 4
Not completed — Lost to Follow-up | 1 | 0 | 1 | 2
Not completed — Lack of Efficacy | 1 | 0 | 1 | 1
Not completed — Other | 1 | 0 | 1 | 0
Not completed — Metformin/Sitagliptin Contraindication | 0 | 0 | 1 | 0
Not completed — Randomized but Not Treated | 0 | 0 | 0 | 1
Not completed — Completion Status Unknown | 1 | 0 | 1 | 0
Period: 80-Week Extension Period
Arm/Group | Placebo | Sitagliptin 100 mg | Fasiglifam 25 mg | Fasiglifam 50 mg
Started | 66 | 138 | 140 | 137
Completed | 0 | 0 | 0 | 0
Not Completed | 66 | 138 | 140 | 137
Not completed — Pregnancy | 0 | 0 | 1 | 0
Not completed — Study Terminated by Sponsor | 65 | 137 | 132 | 132
Not completed — Voluntary Withdrawal | 0 | 1 | 4 | 2
Not completed — Lost to Follow-up | 1 | 0 | 2 | 1
Not completed — Pretreatment Event/Adverse Event | 0 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Sitagliptin 100 mg | Fasiglifam 25 mg | Fasiglifam 50 mg | Total
Number analyzed (Participants) | 132 | 260 | 263 | 261 | 916
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.6 (9.72) | 55.8 (9.84) | 56.3 (9.58) | 56.0 (9.37) | 56.0 (9.60)
Age, Customized [Number; unit: participants]
  < 65 years | 107 | 214 | 216 | 220 | 757
  ≥ 65 years | 25 | 46 | 47 | 41 | 159
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 103 | 127 | 126 | 422
  Male | 66 | 157 | 136 | 135 | 494
Race/Ethnicity, Customized [Number; unit: participants] — Race data is available for 260 participants in the fasiglifam 50 mg treatment arm.
  participants
    American Indian or Alaska Native | 0 | 0 | 2 | 3 | 5
    Asian | 12 | 30 | 28 | 26 | 96
    Black or African American | 8 | 13 | 19 | 12 | 52
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 2 | 2
    White | 112 | 216 | 214 | 217 | 759
    Multiracial | 0 | 1 | 0 | 0 | 1
    Data Not Available | 0 | 0 | 0 | 1 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 13 | 29 | 28 | 28 | 98
  Non-Hispanic or Latino | 28 | 59 | 53 | 55 | 195
  Not Collected | 91 | 172 | 182 | 178 | 623
Region of Enrollment [Number; unit: participants]
  Australia | 3 | 5 | 5 | 5 | 18
  Bulgaria | 3 | 7 | 7 | 7 | 24
  Croatia | 4 | 6 | 8 | 6 | 24
  Czech Republic | 8 | 15 | 14 | 14 | 51
  Hungary | 29 | 56 | 61 | 60 | 206
  Italy | 1 | 3 | 3 | 2 | 9
  Korea, Republic Of | 2 | 4 | 4 | 2 | 12
  Malaysia | 2 | 8 | 7 | 8 | 25
  Slovakia | 34 | 66 | 65 | 66 | 231
  Thailand | 7 | 14 | 13 | 14 | 48
  United States | 39 | 76 | 76 | 77 | 268
Weight [Mean (Standard Deviation); unit: kg] — Weight data is available for 260 participants in the fasiglifam 50 mg treatment arm.
  kg | 91.15 (18.988) | 91.41 (19.664) | 91.44 (17.859) | 91.53 (18.772) | 91.42 (18.776)
Height [Mean (Standard Deviation); unit: cm] — Height data is available for 262 and 260 participants in the fasiglifam 25 mg and fasiglifam 50 mg treatment arms, respectively.
  cm | 168.2 (10.08) | 169.4 (10.74) | 168.5 (10.53) | 168.4 (9.85) | 168.7 (10.34)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI data is available for 262 and 260 participants in the fasiglifam 25 mg and fasiglifam 50 mg treatment arms, respectively.
  kg/m^2 | 32.06 (5.070) | 31.68 (5.282) | 32.11 (5.126) | 32.16 (5.651) | 32.00 (5.312)
BMI Category [Number; unit: participants] — BMI data is available for 262 and 260 participants in the fasiglifam 25 mg and fasiglifam 50 mg treatment arms, respectively.
  participants
    < 30 kg/m^2 | 53 | 106 | 92 | 101 | 352
    ≥ 30 kg/m^2 | 79 | 154 | 170 | 159 | 562
    Data Not Available | 0 | 0 | 1 | 1 | 2
Glycosylated Hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percent] — HbA1c data is available for 258 and 260 participants in the sitagliptin 100 mg and fasiglifam 50 mg treatment arms, respectively.
  percent | 8.34 (0.739) | 8.35 (0.694) | 8.41 (0.712) | 8.43 (0.765) | NA (NA) — Not determined
HbA1c Category [Number; unit: participants] — HbA1c data is available for 260 participants in the fasiglifam 50 mg treatment arm.
  participants
    < 8.5% | 80 | 156 | 154 | 148 | 538
    ≥ 8.5% | 52 | 104 | 109 | 112 | 377
    Data Not Available | 0 | 0 | 0 | 1 | 1
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 6.655 (6.262) | 5.940 (4.942) | 6.726 (4.615) | 6.375 (5.214) | 6.393 (5.143)
Fasting Plasma Glucose [Mean (Standard Deviation); unit: ng/dL] — Data is only available for 258 and 259 participants in the sitagliptin 100 mg and fasiglifam 50 mg treatment arms, respectively.
  ng/dL | 178.4 (36.94) | 175.6 (37.67) | 179.0 (33.52) | 180.0 (37.98) | NA (NA) — Not determined.

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c)
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at Week 24 relative to Baseline. A Mixed Model Repeated Measures (MMRM) model was used for analysis with treatment, country, schedule, visit and visit by treatment interaction as fixed factors and with Baseline value and Baseline value by visit interaction as covariates with an unstructured covariance structure.
Time Frame: Baseline and Week 24
Population: Full Analysis Set included all randomized participants who received at least 1 dose of study drug analyzed according to the treatment group to which they were randomized. A participant was included in the analyses when there was both a Baseline and at least 1 Post-baseline value at Week 24.
Measure: Least Squares Mean (Standard Error); unit: Percent
Arm/Group | Placebo | Sitagliptin 100 mg | Fasiglifam 25 mg | Fasiglifam 50 mg
Number analyzed (Participants) | 67 | 145 | 144 | 138
Percent | -0.19 (0.098) | -1.07 (0.074) | -0.75 (0.073) | -1.01 (0.074)
Statistical Analysis 1: Comparison: Placebo vs Fasiglifam 25 mg; Test type: Superiority or Other; p < 0.001, Mixed model for repeated measurements — MMRM model with treatment, country, schedule, visit and visit by treatment interaction as fixed factors and with baseline value and baseline value by visit interaction as covariates with an unstructured covariance structure; LS Mean Difference = -0.55, 95% CI 2-sided [-0.77 to -0.34], Standard Error of Mean 0.108
Statistical Analysis 2: Comparison: Sitagliptin 100 mg vs Fasiglifam 25 mg; Test type: Superiority or Other; p < 0.001, Mixed model for repeated measurements — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = 0.32, 95% CI 2-sided [0.15 to 0.49], Standard Error of Mean 0.087
Statistical Analysis 3: Comparison: Placebo vs Fasiglifam 50 mg; Test type: Superiority or Other; p < 0.001, Mixed model for repeated measurements — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -0.82, 95% CI 2-sided [-1.03 to -0.60], Standard Error of Mean 0.109
Statistical Analysis 4: Comparison: Sitagliptin 100 mg vs Fasiglifam 50 mg; Test type: Superiority or Other; p = 0.524, Mixed model for repeated measurements — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = 0.06, 95% CI 2-sided [-0.12 to 0.23], Standard Error of Mean 0.087

2. Secondary Outcome: Incidence of HbA1c <7%
Description: Incidence (percentage) of participants with glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) less than 7% at Week 24.
Time Frame: 24 Weeks
Population: Full Analysis Set included all randomized participants who received at least 1 dose of study drug analyzed according to the treatment group to which they were randomized
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Sitagliptin 100 mg | Fasiglifam 25 mg | Fasiglifam 50 mg
Number analyzed (Participants) | 67 | 145 | 144 | 138
percentage of participants | 14.9 | 42.8 | 24.3 | 37.0
Statistical Analysis 1: Comparison: Placebo vs Fasiglifam 25 mg; Test type: Superiority or Other; p = 0.050, Regression, Logistic — P-Value was obtained from a logistic model with treatment, schedule, baseline HbA1c as explanatory variables; Odds Ratio (OR) = 2.25, 95% CI 2-sided [1.00 to 5.08]
Statistical Analysis 2: Comparison: Sitagliptin 100 mg vs Fasiglifam 25 mg; Test type: Superiority or Other; p < 0.001, Regression, Logistic — P-Value was obtained from a logistic model with treatment, schedule, baseline HbA1c as explanatory variables; Odds Ratio (OR) = 0.39, 95% CI 2-sided [0.23 to 0.67]
Statistical Analysis 3: Comparison: Placebo vs Fasiglifam 50 mg; Test type: Superiority or Other; p < 0.001, Regression, Logistic — P-Value was obtained from a logistic model with treatment, schedule, baseline HbA1c as explanatory variables; Odds Ratio (OR) = 5.06, 95% CI 2-sided [2.24 to 11.42]
Statistical Analysis 4: Comparison: Sitagliptin 100 mg vs Fasiglifam 50 mg; Test type: Superiority or Other; p = 0.493, Regression, Logistic — P-Value was obtained from a logistic model with treatment, schedule, baseline HbA1c as explanatory variables; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.50 to 1.39]

3. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG)
Description: The change between FPG collected at week 24 relative to Baseline. A MMRM model was used for analysis with treatment, country, schedule, visit and visit by treatment interaction as fixed factors and with Baseline value and Baseline value by visit interaction as covariates with an unstructured covariance structure.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Sitagliptin 100 mg | Fasiglifam 25 mg | Fasiglifam 50 mg
Number analyzed (Participants) | 67 | 145 | 142 | 135
mg/dL | -1.6 (4.07) | -21.7 (3.13) | -26.9 (3.13) | -32.9 (3.18)
Statistical Analysis 1: Comparison: Placebo vs Fasiglifam 25 mg; Test type: Superiority or Other; p < 0.001, Mixed model for repeated measurements — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -25.2, 95% CI 2-sided [-33.8 to -16.6], Standard Error of Mean 4.36
Statistical Analysis 2: Comparison: Sitagliptin 100 mg vs Fasiglifam 25 mg; Test type: Superiority or Other; p = 0.142, Mixed model for repeated measurements — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -5.1, 95% CI 2-sided [-12.0 to 1.7], Standard Error of Mean 3.49
Statistical Analysis 3: Comparison: Placebo vs Fasiglifam 50 mg; Test type: Superiority or Other; p < 0.001, Mixed model for repeated measurements — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -31.3, 95% CI 2-sided [-39.9 to -22.6], Standard Error of Mean 4.40
Statistical Analysis 4: Comparison: Sitagliptin 100 mg vs Fasiglifam 50 mg; Test type: Superiority or Other; p = 0.002, Mixed model for repeated measurements — [p-value comment as in outcome 1, analysis 1]; Least Square Mean difference = -11.2, 95% CI 2-sided [-18.1 to -4.2], Standard Error of Mean 3.53

ADVERSE EVENTS:
Time Frame: First dose of study medication to 30 day past last dose of study medication (Up to 637 days)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Placebo | Sitagliptin 100 mg | Fasiglifam 25 mg | Fasiglifam 50 mg
Serious Adverse Events (participants affected / at risk) | 2/132 | 10/260 | 14/263 | 4/260
Other Adverse Events (participants affected / at risk) | 17/132 | 16/260 | 18/263 | 20/260
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=132) | Sitagliptin 100 mg (N=260) | Fasiglifam 25 mg (N=263) | Fasiglifam 50 mg (N=260)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 1 | 0
Phimosis (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Gangrene (Infections and infestations) | 0 | 0 | 1 | 0
Hepatitis B (Infections and infestations) | 0 | 1 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 2 | 0 | 0 — One treatment-emergent death occurred during treatment with sitagliptin and is not related.
Erysipelas (Infections and infestations) | 0 | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 1 | 0 | 0
Carotid bruit (Investigations) | 0 | 1 | 0 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Tumour of ampulla of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 — One treatment-emergent death occurred during treatment with placebo and is not related.
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Radiculopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 1 | 0 | 0
Peripheral artery stenosis (Vascular disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=132) | Sitagliptin 100 mg (N=260) | Fasiglifam 25 mg (N=263) | Fasiglifam 50 mg (N=260)
Hyperglycaemia (Metabolism and nutrition disorders) | 14 | 9 | 11 | 7
Nasopharyngitis (Infections and infestations) | 3 | 8 | 7 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.